CLINICAL TRIAL: NCT07207850
Title: Parents Helping Parents for Youth Vaping Cessation (PhP-VX)
Brief Title: Parents Helping Parents for Youth Vaping Cessation
Acronym: PhP-VX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Massachusetts General Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hongying Daisy Dai, Principal Investigator, University of Nebraska
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0617-25-EP; 1R34CA287719-01A1 (NIH)
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Implementation Science; Engagement, Patient; E Cigarette Use; Peer Support; Vaping Teens; Vaping Cessation; Parent Support
Keywords: Vaping; Tobacco; vaping cessation; Parent support; adolescent vaping
MeSH Terms: conditions — Patient Participation; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in this arm will not receive the PhP-VX treatment.
- Test Group - PHP-VX Program (Experimental): Participants in this arm will receive the PhP-VX program.
  Interventions: Behavioral: Parents Helping Parents program

INTERVENTIONS:
Behavioral: Parents Helping Parents program — Our innovative vaping cessation program will include two key components: 1) online training for parents and their offspring, and 2) parent-helping-parent coach sessions. Parents and children in the control setting will receive no treatments during the intervention (Baseline to Month 3). Dyads will be provided online training materials after the 6 month follow up.
  Arms: Test Group - PHP-VX Program

SUMMARY:
The goal of this randomized controlled study is to test if this new intervention works to help adolescents quit vaping. A key feature of the program is the use of peer support for parents, delivered by trained parent coaches. Participants will complete baseline and follow up surveys. Parents in the intervention arm will receive peer support as part of the program.

DETAILED DESCRIPTION:
This objective of study is to develop and test the feasibility of a novel Parents-helping-Parents for Youth Vaping Cessation (PhP-VX) program. The investigators will conduct a feasibility pilot test with 100 parent-adolescent dyads recruited from an EHR system. Half of the dyads will receive the "PhP-VX" program for 3 months, and half of the dyads will be assigned to the control (no-treatment) group.

The PhP-VX program consists of two key components: 1) online lessons for participating parents and adolescents and 2) one on one sessions with a coach for parents.

Eligible dyads will be randomly assigned to either the test or control group using a computer-generated randomization list. At baseline, all participants will complete a survey assessing their e-cigarette and tobacco use, vaping knowledge, and exposure to marketing and media. Dyads assigned to the test arm will receive PhP-VX program instructions, and parents will be immediately connected with a coach. Parents will be scheduled to receive six bi-weekly, 30-minute, 1:1 coach-facilitated sessions via Zoom. The coaches will identify the priority needs of the participant, provide support and advocacy (e.g., coach on how to identify own needs and access resources), role model (e.g., share experiences, demonstrate effective decision-making), effective communication with their children, and facilitate change (motivation, facilitate change through goal setting/education/skills building). Parents will also be able to contact the coach as needed for additional support and resources.

All participants in both the control and test arms will be followed up at months 1, 3, and 6 with questions on e-cigarette use, vaping knowledge, and marketing/media literacy. Parents and children in the test arm will also complete an evaluation of the PhP-VX program at the end of the intervention (month 3).

The investigators will offer twenty adolescent participants (10 control, 10 intervention) the option to provide saliva samples at baseline, 3 months, and 6 months. The samples will be collected using the iScreen Oral Fluid Device (OFD) cotinine test, which detects cotinine, a metabolite of nicotine and the recommended biomarker for validating self-reported tobacco abstinence. Cotinine levels will serve as our biochemical verification of participants' self-reported abstinence. Adolescents who agree to participate will receive saliva collection kits by mail. Participants will be instructed to upload a photo of their test result via a REDCap survey.

Parents and children in the control group, who receive no intervention during the study, will be given access to online training materials following the final follow-up at month 6.

ELIGIBILITY:
ADOLESCENT INCLUSION:

* 15-18
* Report vaping in the previous 30 days
* English literacy

PARENT INCLUSION:

* Biological, adoptive, stepparents, or adult guardian of adolescent participating
* Have face-to-face contact with the adolescent at least one day per week during the study period
* Access to a computer or mobile phone at home
* Interested in helping adolescent quit e-cigarette/vape use

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence abstinence | Baseline and Follow ups (1 month, 3 months, 6 months)

SECONDARY OUTCOMES:
Vaping frequency | Baseline and Follow ups (1 month, 3 months, 6 months)
Past 7 day Vaping intensity | Baseline and Follow ups (1 month, 3 months, 6 months)
  Self-reported vaping intensity will be assessed with the questions "In the past 7 days, on the days you vaped, how many times did you usually pick up your device to vape? "and "In the past 7 days, each time you pick up your vape, how many puffs do you usually take before putting it away?".
Other tobacco use | Baseline and Follow ups (1 month, 3 months, 6 months)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual, aggregated, summarized data will be made available for sharing. To facilitate interpretation of the data, statistical analysis plans will be created, shared, and associated with the relevant datasets.
Supporting Information: SAP
Time Frame: Shared data generated from this project will be made available upon publications. The duration of preservation and sharing of the data will be a minimum of 10 years after the end of the funding period.
Access Criteria: Summary information on the data shared in NDA is available in the NDA Query Tool without the need for an NDA user account. To request access to record-level human subject data, you must submit a Data Access Request.
URL: https://nda.nih.gov/